CLINICAL TRIAL: NCT02652260
Title: Phase IIb, Double-Blinded, Multicenter, Randomized Study to Assess the Effect on Central Nervous System (CNS) Toxicity of Switching From ATRIPLA™ (Efavirenz, Tenofovir, Emtricitabine) to MK-1439A (Doravirine, Tenofovir, Lamivudine) in Virologically-Suppressed Subjects.
Brief Title: Effects of Switching From ATRIPLA™ (Efavirenz, Tenofovir, Emtricitabine) to MK-1439A (Doravirine, Tenofovir, Lamivudine) in Virologically-Suppressed Participants (MK-1439A-028)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1439A-028; MK-1439A-028 (Other: Merck Protocol Number); 2015-003617-18 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: HIV-1; Central Nervous System
MeSH Terms: interventions — doravirine; Tenofovir; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Switch to Doravirine, Tenofovir, Lamivudine (Experimental): Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening will be switched to blinded doravirine, tenofovir, lamivudine orally, once daily for 12 weeks, followed by open-label doravirine, tenofovir, lamivudine orally, once daily for an additional 12 weeks. Participants who meet eligibility criteria can enter study extension 1 to receive open-label doravirine, tenofovir, lamivudine for an additional 96 weeks. Participants who meet eligibility criteria can enter study extension 2 to receive open-label doravirine, tenofovir, lamivudine, with a maximum total duration of treatment of 216 weeks. Participants who meet eligibility criteria can enter study extension 3 to receive open-label doravirine, tenofovir, lamivudine, with a maximum total duration of treatment of 312 weeks.
  Interventions: Drug: Doravirine, Tenofovir, Lamivudine - Blinded; Drug: Doravirine, Tenofovir, Lamivudine - Open-Label; Drug: Placebo to ATRIPLA™
- Deferred Switch to Doravirine, Tenofovir, Lamivudine (Experimental): Participants will continue on their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks, followed by open-label doravirine, tenofovir, lamivudine orally, once daily for 24 weeks. Participants who meet eligibility criteria can enter study extension 1 to receive open-label doravirine, tenofovir, lamivudine for an additional 96 weeks. Participants who meet eligibility criteria can enter study extension 2 to receive open-label doravirine, tenofovir, lamivudine, with a maximum total duration of treatment of 228 weeks. Participants who meet eligibility criteria can enter study extension 3 to receive open-label doravirine, tenofovir, lamivudine, with a maximum total duration of treatment of 324 weeks.
  Interventions: Drug: Doravirine, Tenofovir, Lamivudine - Open-Label; Drug: ATRIPLA^TM; Drug: Placebo to Doravirine, Tenofovir, Lamivudine

INTERVENTIONS:
Drug: Doravirine, Tenofovir, Lamivudine - Blinded — A single tablet FDC containing doravirine 100 mg, lamivudine (3TC) 300 mg and tenofovir disoproxil fumarate (TDF) 300 mg administered orally, once daily for 12 weeks during the Blinded period
  Other Names: MK-1439A
  Arms: Immediate Switch to Doravirine, Tenofovir, Lamivudine
Drug: Doravirine, Tenofovir, Lamivudine - Open-Label — A single-tablet FDC containing doravirine 100 mg, 3TC 300 mg and TDF 300 mg administered orally, once daily for either 12 or 24 weeks during the Open-Label Period; also an additional 96 weeks during the Open-Label extension period 1; a maximum total duration of treatment of 228 weeks during the Open-Label extension period 2; and a maximum total duration of treatment of 324 weeks during the Open-Label extension period 3.
  Other Names: MK-1439A
Drug: ATRIPLA^TM — A single tablet FDC containing efavirenz (EFV) 600 mg, emtricitabine (FTC) 200 mg, and TDF 300 mg administered orally, once daily for 12 weeks during the Blinded period
  Arms: Deferred Switch to Doravirine, Tenofovir, Lamivudine
Drug: Placebo to ATRIPLA™ — A single placebo to ATRIPLA™ tablet administered orally, once daily for 12 weeks during the Blinded period
  Arms: Immediate Switch to Doravirine, Tenofovir, Lamivudine
Drug: Placebo to Doravirine, Tenofovir, Lamivudine — A single placebo to doravirine, tenofovir, lamivudine tablet administered orally, once daily for 12 weeks during the Blinded period
  Arms: Deferred Switch to Doravirine, Tenofovir, Lamivudine

SUMMARY:
This study aims to evaluate a switch from fixed dose combination (FDC) treatment with ATRIPLA^TM for 12 weeks prior to screening to FDC treatment with Doravirine, Tenofovir, Lamivudine (MK-1439A) in virologically-suppressed, human immunodeficiency virus type 1 (HIV-1)-infected participants. The primary hypothesis is that switching from ATRIPLA^TM to Doravirine, Tenofovir, Lamivudine results in a lower proportion of participants with at least one CNS toxicity of at least Grade 2 intensity at Week 12 than continuation of ATRIPLA^TM treatment.

ELIGIBILITY:
Inclusion Criteria:

* is taking ATRIPLA™, generic versions of ATRIPLA™, or the components of ATRIPLA™ (EFV,TDF plus emtricitabine),
* has documentation of HIV-1 ribonucleic acid (RNA) < 50 copies/mL during the 12 weeks prior to screening while on ATRIPLA™.
* has plasma HIV-1 RNA levels below the limits of quantification (BLoQ) at the screening visit.
* if genotyped prior to starting initial antiretroviral regimen, must have no known resistance to any of the study agents
* has at least one EFV-associated CNS toxicities of Grade 2 or worse intensity both at the time of screening and at Study Day 1
* is highly unlikely to become pregnant or to impregnate a partner
* To be eligible for study extension 1, participants from Immediate Switch Group (ISG) must have completed Study Week 24, and benefited from study participation; participants from Deferred Switch Group (DSG) must have completed Study Week 36, and benefited from study participation as determined by the investigator
* To be eligible for study extension 2, participants from ISG must have completed Study Week 120, and benefited from study participation; participants from DSG must have completed Study Week 132, and benefited from study participation as determined by the investigator

Exclusion Criteria:

* is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.
* has ongoing Grade 4 CNS toxicity during screening period that requires a prompt change in ART
* has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1 including, but not limited to, adefovir, emtricitabine, entecavir, lamivudine or tenofovir.
* has documented or known resistance to study drugs including doravirine, lamivudine, and/or tenofovir
* has participated in, or anticipates participating in a study with an investigational compound/device within 30 days prior to signing informed consent
* has used systemic immunosuppressive therapy or immune modulators or anticipates using them within 30 days prior to this study
* requires or anticipates requiring any of the prohibited medications
* has significant hypersensitivity or other contraindication to any of the components of the study drugs
* has a current (active) diagnosis of acute hepatitis due to any cause.
* has evidence of decompensated liver disease manifested by the presence of or a history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver diseases, or has liver cirrhosis and a Child-Pugh Class C score or Pugh-Turcotte (CPT) score > 9.
* is pregnant, breastfeeding, or expecting to conceive.
* female is expecting to donate eggs (at any time during the study) or male is expecting to donate sperm (at any time during the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Nelson M, Winston A, Hill A, Mngqibisa R, Bassa A, Orkin C, Rassool M, Rodgers A, Teal V, Kumar S, Teppler H. Efficacy, safety and central nervous system effects after switch from efavirenz/tenofovir/emtricitabine to doravirine/tenofovir/lamivudine. AIDS. 2021 Apr 1;35(5):759-767. doi: 10.1097/QAD.0000000000002804. PMID 33587439
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 112 participants screened, 86 were randomized and received study treatment.
Groups:
- Immediate Switch to MK-1439A: Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening were switched to blinded MK-1439A orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for an additional 12 weeks. Eligible participants from Base Study (Day 1 to Week 24) may have entered open-label optional study extensions to receive MK-1439A once daily during Study Extension 1 (Weeks 24 to 120), Extension 2 (Weeks 120 to 216), and Extension 3 (Weeks 216 to 312).
- Deferred Switch to MK-1439A: Participants continued their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks (Day 1 to Week 12), followed by open-label MK-1439A orally, once daily for 24 weeks (Weeks 12 to 36). Eligible participants from Base Study (Day 1 to Week 36) may have entered open-label optional study extensions to receive MK-1439A once daily during Study Extension 1 (Weeks 36 to 132), Extension 2 (Weeks 132 to 228), and Extension 3 (Weeks 228 to 324).
Period: Base Study
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Started | 43 | 43
Switched Over to MK-1439A | 0 | 42
Completed | 43 | 41
Not Completed | 0 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Study Extension 1 (Open-Label)
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Started | 43 | 41
Completed | 39 | 34
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Pregnancy | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Availability of study drug locally | 1 | 1
Not completed — Adverse Event | 0 | 2
Period: Study Extension 2 (Open-Label)
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Started (Not all study participants continued into optional study extension 2) | 39 | 33
Completed | 17 | 19
Not Completed | 22 | 14
Not completed — Adverse Event | 1 | 0
Not completed — Availability of study drug locally | 18 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-Compliance with study drug | 1 | 0
Not completed — Pregnancy | 1 | 1
Period: Study Extension 3 (Open-Label)
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Started | 17 | 19
Completed | 10 | 8
Not Completed | 7 | 11
Not completed — Physician Decision | 7 | 10
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Immediate Switch to MK-1439A: Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening will be switched to blinded MK-1439A orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for an additional 12 weeks. Eligible participants from Base Study (Day 1 to Week 24) may have entered open-label optional study extensions to receive MK-1439A once daily during Study Extension 1 (Weeks 24 to 120), Extension 2 (Weeks 120 to 216), and Extension 3 (Weeks 216 to 312).
- Total: Total of all reporting groups
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (11.9) | 41.6 (11.2) | 41.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 39 | 42 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 23 | 48
  White | 12 | 19 | 31
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
CNS Toxicity Percentage Of Maximum Score [Mean (Standard Deviation); unit: Percentage of maximum score] — Participants were asked to rate the intensity for each of the 10 events as none (Grade 0), mild (Grade 1), moderate (Grade 2), or severe (Grade 3). Mild = symptom is noticeable but does not interfere with normal activities; moderate = symptom has some impact on normal activities; severe = symptom prevents conduct of normal activities. The CNS toxicity score was calculated by summing across all 10 CNS toxicities and converting the sum to a percentage of the maximum possible sum of intensities (10 x 3 = 30). A higher CNS score indicates worsening symptoms.
  Percentage of maximum score | 32.9 (16.5) | 37.1 (19.0) | 35.0 (17.8)
Fasting Lipids [Mean (Standard Deviation); unit: mg/dL] — Mean concentrations of low-density lipoprotein (LDL) cholesterol; Non high-density lipoprotein (HDL) cholesterol; cholesterol; HDL cholesterol; and triglyceride. Population: All randomized participants who received at least one dose of study treatment.
  mg/dL
    LDL Cholesterol: number analyzed (Participants) | 36 | 41 | 77
    LDL Cholesterol | 98.67 (35.28) | 99.54 (33.57) | 99.13 (34.15)
    Non-HDL Cholesterol: number analyzed (Participants) | 37 | 41 | 78
    Non-HDL Cholesterol | 118.73 (36.93) | 117.76 (37.83) | 118.22 (37.16)
    Cholesterol: number analyzed (Participants) | 37 | 41 | 78
    Cholesterol | 178.11 (36.39) | 173.02 (36.62) | 175.44 (36.37)
    HDL Cholesterol: number analyzed (Participants) | 37 | 41 | 78
    HDL Cholesterol | 59.38 (14.58) | 55.27 (14.00) | 57.22 (14.34)
    Triglyceride: number analyzed (Participants) | 37 | 41 | 78
    Triglyceride | 107.49 (65.64) | 91.39 (39.43) | 99.03 (53.73)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Central Nervous System (CNS) Toxicity of at Least Grade 2 Intensity at Week 12
Description: A questionnaire was used to solicit for CNS toxicity based on the following 10 events: dizziness; depression/low mood; insomnia/sleeplessness; anxiety/nervousness; confusion; impaired concentration/attention; headache; somnolence/daytime sleepiness; aggressive mood/behavior; and abnormal dreams. Participants were asked to rate the intensity for each of the 10 events as none (Grade 0), mild (Grade 1), moderate (Grade 2), or severe (Grade 3). Mild = symptom is noticeable but does not interfere with normal activities; moderate = symptom has some impact on normal activities; severe = symptom prevents conduct of normal activities. Percentage of participants with at least one CNS toxicity of Grade 2 or higher were recorded, based on the last observation carried forward (LOCF) approach.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study treatment, and have baseline data for analyses requiring baseline data.
Measure: Number; unit: Percentage of participants
Groups:
- Immediate Switch to MK-1439A: Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening will be switched to blinded MK-1439A orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for an additional 12 weeks.
- Deferred Switch to MK-1439A: Participants will continue on their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for 24 weeks.
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Percentage of participants | 41.9 | 37.2
Statistical Analysis 1: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Treatment Difference: Immediate Switch minus Delayed Switch; Test type: Other — The Immediate Switch group will be considered statistically significantly smaller than the Delayed Switch group if the upper bound of the 95% confidence interval for the treatment difference is less than 0; p = 0.331, Miettinen and Nurminen; Estimated Difference = 4.65, 95% CI 2-sided [-15.92 to 24.85]; The 95% confidence interval (CI) was calculated by the method of Miettinen and Nurminen

2. Secondary Outcome: Percentage of Participants With at Least One CNS Toxicity of at Least Grade 2 Intensity at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Percentage of participants | 46.5 | 65.1
Statistical Analysis 1: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Treatment Difference: Immediate Switch minus Delayed Switch; Test type: Other — [test comment as in outcome 1, analysis 1]; Estimated Difference = -18.61, 95% CI 2-sided [-38.14 to 2.51]; The 95% CI was calculated by the method of Miettinen and Nurminen

3. Secondary Outcome: Change From Baseline in CNS Toxicity Score at Week 4
Description: A questionnaire was used to solicit for CNS toxicity based on the following 10 events: dizziness; depression/low mood; insomnia/sleeplessness; anxiety/nervousness; confusion; impaired concentration/attention; headache; somnolence/daytime sleepiness; aggressive mood/behavior; and abnormal dreams. Participants were asked to rate the intensity for each of the 10 events as none (Grade 0), mild (Grade 1), moderate (Grade 2), or severe (Grade 3). Mild = symptom is noticeable but does not interfere with normal activities; moderate = symptom has some impact on normal activities; severe = symptom prevents conduct of normal activities. The CNS toxicity score was calculated by summing across all 10 CNS toxicities and converting the sum to a percentage of the maximum possible sum of intensities (10 x 3 = 30). A positive change from baseline score indicates worsening symptoms. A negative change from baseline score indicates improvement in symptoms.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of maximum score
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Percentage of maximum score | -17.6 [-23.4 to -11.8] | -15.6 [-22.0 to -9.2]
Statistical Analysis 1: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Treatment Difference: Immediate Switch minus Delayed Switch; Test type: Other; Estimated Difference = -2.0, 95% CI 2-sided [-10.5 to 6.5]; The 95% CI was based on a t-distribution

4. Secondary Outcome: Change From Baseline in CNS Toxicity Score at Week 12
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of maximum score
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Percentage of maximum score | -18.1 [-22.9 to -13.3] | -21.7 [-27.9 to -15.5]
Statistical Analysis 1: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Treatment Difference: Immediate Switch minus Delayed Switch; Test type: Other; Estimated Difference = 3.6, 95% CI 2-sided [-4.1 to 11.3]; The 95% CI was calculated by the method of Miettinen and Nurminen

5. Secondary Outcome: Percentage of Participants With at Least One CNS Toxicity of at Least Grade 2 Intensity at Time of Switch, and at 24 Weeks Post-switch for the Combined Treatment Groups
Description: A questionnaire was used to solicit for CNS toxicity based on the following 10 events: dizziness; depression/low mood; insomnia/sleeplessness; anxiety/nervousness; confusion; impaired concentration/attention; headache; somnolence/daytime sleepiness; aggressive mood/behavior; and abnormal dreams. Participants were asked to rate the intensity for each of the 10 events as none (Grade 0), mild (Grade 1), moderate (Grade 2), or severe (Grade 3). Mild = symptom is noticeable but does not interfere with normal activities; moderate = symptom has some impact on normal activities; severe = symptom prevents conduct of normal activities. For the Immediate Switch Group (ISG) time of switch was study Day 1, and week 24 post-switch was week 24. For the Delayed Switch Group (DSG) time of switch was study week 12, and week 24 post-switch was week 36.
Time Frame: Baseline (time of switch) and 24 weeks post-switch
Population: All randomized participants who received at least one dose of study treatment, and have baseline data for analyses requiring baseline data. Based on the protocol-specified plan, the combined treatment groups was analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- Combined Treatment Groups: Time of Switch; Combined Treatment Groups: Week 24 Post-Switch: Immediate Switch to MK-1439A: Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening will be switched to blinded MK-1439A orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for an additional 12 weeks.
  Deferred Switch to MK-1439A: Participants will continue on their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for 24 weeks.
Arm/Group | Combined Treatment Groups: Time of Switch | Combined Treatment Groups: Week 24 Post-Switch
Number analyzed (Participants) | 86 | 86
Percentage of participants | 68.6 | 30.2
Statistical Analysis 1: Comparison: Combined Treatment Groups: Time of Switch vs Combined Treatment Groups: Week 24 Post-Switch; Change from time of switch to 24 weeks post-switch: Treatment difference in percent response; Test type: Other — The 95% CI was calculated by the method of Miettinen and Nurminen; Difference in Percentage = -38.4, 95% CI 2-sided [-51.2 to -23.8]; Week 24 Post-switch minus Time of switch

6. Secondary Outcome: CNS Toxicity Scores at Time of Switch, and at 24 Weeks Post-switch for the Combined Treatment Groups
Description: A questionnaire was used to solicit for CNS toxicity based on the following 10 events: dizziness; depression/low mood; insomnia/sleeplessness; anxiety/nervousness; confusion; impaired concentration/attention; headache; somnolence/daytime sleepiness; aggressive mood/behavior; and abnormal dreams. Participants were asked to rate the intensity for each of the 10 events as none (Grade 0), mild (Grade 1), moderate (Grade 2), or severe (Grade 3). The CNS toxicity score was calculated by summing across all 10 CNS toxicities and converting the sum to a percentage of the maximum possible sum of intensities (10 x 3 = 30). A higher CNS score indicates worse symptoms. A positive change in CNS score indicates worsening symptoms. A negative change indicates improvement in symptoms. For the ISG time of switch was study Day 1, and week 24 post-switch was week 24. For the DSG time of switch was study week 12, and week 24 post-switch was week 36.
Time Frame: Baseline (time of switch) and 24 weeks post-switch
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Percentage of maximum score
Arm/Group | Combined Treatment Groups: Time of Switch | Combined Treatment Groups: Week 24 Post-Switch
Number analyzed (Participants) | 86 | 86
Percentage of maximum score | 24.2 [20.5 to 27.9] | 10.7 [8.7 to 12.8]
Statistical Analysis 1: Comparison: Combined Treatment Groups: Time of Switch vs Combined Treatment Groups: Week 24 Post-Switch; Change from time of switch to 24 weeks post-switch: Treatment difference in score; Test type: Other — The 95% CI was based on a t-distribution; Mean Difference (Final Values) = -13.4, 95% CI 2-sided [-16.8 to -10.1]; Week 24 Post-switch minus Time of switch

7. Secondary Outcome: Change From Baseline in Fasting Lipids at Week 12
Description: Blood was collected under fasting conditions on Day 1 and on week 12 in order to determine the concentration of the following lipids: low-density lipoprotein (LDL) cholesterol; Non high-density lipoprotein (HDL) cholesterol; cholesterol; HDL cholesterol; and triglyceride.
Time Frame: Baseline (study Day 1) and study week 12
Population: All randomized participants who received at least one dose of study treatment, and have required lipid data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 37 | 41
mg/dL
  LDL Cholesterol: number analyzed (Participants) | 36 | 41
  LDL Cholesterol | -10.78 (15.85) | -1.88 (14.88)
  Non-HDL Cholesterol | -14.08 (17.17) | -0.37 (16.51)
  Cholesterol | -22.14 (19.49) | 0.00 (18.04)
  HDL Cholesterol | -8.05 (7.74) | 0.37 (7.91)
  Triglyceride | -21.19 (43.37) | 7.10 (38.55)
Statistical Analysis 1: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Difference Estimate: LDL Cholesterol; Test type: Other — The 95% CI for treatment difference was calculated from an ANCOVA model with terms for baseline lipid level, use of lipid lowering therapy at study Day 1 and treatment; Difference Estimate = -9.02, 95% CI 2-sided [-15.69 to -2.35]; ISG minus DSG
Statistical Analysis 2: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Difference Estimate: Non-HDL Cholesterol; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference Estimate = -13.57, 95% CI 2-sided [-20.79 to -6.35]; ISG minus DSG
Statistical Analysis 3: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Difference Estimate: Cholesterol; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference Estimate = -21.42, 95% CI 2-sided [-29.63 to -13.21]; ISG minus DSG
Statistical Analysis 4: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Difference Estimate: HDL Cholesterol; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference Estimate = -8.18, 95% CI 2-sided [-11.76 to -4.60]; ISG minus DSG
Statistical Analysis 5: Comparison: Immediate Switch to MK-1439A vs Deferred Switch to MK-1439A; Difference Estimate: Triglyceride; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference Estimate = -22.18, 95% CI 2-sided [-38.52 to -5.84]; ISG minus DSG

8. Secondary Outcome: Change in Fasting Lipids Between Time of Switch and Week 24 Post-switch for the Combined Treatment Groups
Description: Blood was collected under fasting conditions at time of switch and 24 weeks post-switch in order to determine the change from baseline of the following lipids: low-density lipoprotein (LDL) cholesterol; Non high-density lipoprotein (HDL) cholesterol; cholesterol; HDL cholesterol; and triglyceride. For the ISG time of switch was study Day 1, and week 24 post-switch was week 24. For the DSG time of switch was study week 12, and week 24 post-switch was week 36.
Time Frame: Baseline (time of switch) and 24 weeks post-switch
Population: All randomized participants who received at least one dose of study treatment, and have required lipid data. Based on the protocol-specified plan, the combined treatment groups was analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Combined Treatment Groups: Immediate Switch to MK-1439A: Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening will be switched to blinded MK-1439A orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for an additional 12 weeks.
  Deferred Switch to MK-1439A: Participants will continue on their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks, followed by open-label MK-1439A orally, once daily for 24 weeks.
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 76
mg/dL
  LDL Cholesterol: number analyzed (Participants) | 75
  LDL Cholesterol | -10.97 (17.15)
  Non-HDL Cholesterol | -13.18 (19.82)
  Cholesterol | -20.91 (20.19)
  HDL Cholesterol | -7.72 (9.53)
  Triglyceride | -12.99 (46.61)

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 and <40 Copies/ml at Week 24 Post-switch for the Combined Treatment Groups
Description: Blood was collected under fasting conditions at 24 weeks post-switch in order to determine the HIV-1 RNA. For the ISG week 24 post-switch was week 24. For the DSG week 24 post-switch was week 36.
Time Frame: 24 weeks post-switch
Population: All randomized participants who received at least one dose of study treatment, and have required HIV-1 RNA data. Based on the protocol-specified plan, the combined treatment groups was analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Percentage of participants
  < 50 copies/mL | 95.3 [88.4 to 98.7]
  < 40 copies/mL | 95.3 [88.4 to 98.7]

10. Secondary Outcome: Change From Time of Switch to Week 24 Post Switch in CD4 T-cell Count for the Combined Treatment Groups
Description: Blood was collected at time of switch and at 24 weeks post-switch in order to determine the CD4 T-cell count. For the ISG time of switch was study Day 1, and week 24 post-switch was week 24. For the DSG time of switch was study week 12, and week 24 post-switch was week 36.
Time Frame: Baseline (time of switch) and 24 weeks post-switch
Population: All randomized participants who received at least one dose of study treatment, and have required CD4 T-cell data. Based on the protocol-specified plan, the combined treatment groups was analyzed.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
cells/mm^3 | 70.4 [35.9 to 104.8]

11. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs) Through Study Week 12
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 12
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Participants | 34 | 34

12. Secondary Outcome: Number of Participants With One or More Drug-related AEs Through Study Week 12
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. A drug-related AE was determined by the investigator to be related to the drug.
Time Frame: Up to Week 12
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Participants | 14 | 9

13. Secondary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs) Through Study Week 12
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that results in any of the following: death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; is associated with an overdose.
Time Frame: Up to Week 12
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With One or More Drug-related SAEs Through Study Week 12
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that results in any of the following: death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; is associated with an overdose. A drug-related SAE was determined by the investigator to be related to the drug.
Time Frame: Up to Week 12
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

15. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to an AE Through Study Week 12
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 12
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Switch to MK-1439A | Deferred Switch to MK-1439A
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With One or More AEs for the Combined Treatment Groups 24 Weeks After the Switch
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. For the ISG 24 week post-switch was week 24; for the DSG week 24 post-switch was week 36.
Time Frame: 24 weeks post-switch
Population: All randomized participants who received at least one dose of study treatment, and have baseline data for analyses requiring baseline data. Based on the protocol-specified plan, the combined treatment groups was analyzed. One participant in the DSG who discontinued from the study, before switching to MK-1439A, was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Participants | 71

17. Secondary Outcome: Number of Participants With One or More Drug-related AEs for the Combined Treatment Groups 24 Weeks After the Switch
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol - specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. A drug-related AE was determined by the investigator to be related to the drug. For the ISG 24 week post-switch was week 24; for the DSG week 24 post-switch was week 36.
Time Frame: 24 weeks post-switch
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Participants | 18

18. Secondary Outcome: Number of Participants With One or More SAEs for the Combined Treatment Groups 24 Weeks After the Switch
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that results in any of the following: death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; is associated with an overdose. For the ISG 24 week post-switch was week 24; for the DSG week 24 post-switch was week 36.
Time Frame: 24 weeks post-switch
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Participants | 1

19. Secondary Outcome: Number of Participants With One or More Drug-related SAEs for the Combined Treatment Groups 24 Weeks After the Switch
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that results in any of the following: death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; is associated with an overdose. A drug-related SAE was determined by the investigator to be related to the drug. For the ISG 24 week post-switch was week 24; for the DSG week 24 post-switch was week 36.
Time Frame: 24 weeks post-switch
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Participants | 0

20. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to an AE for the Combined Treatment Groups 24 Weeks After the Switch
Description: as for outcome 16
Time Frame: 24 weeks post-switch
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Groups
Number analyzed (Participants) | 85
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 326 weeks
Description: All cause-mortality was reported on all allocated participants. Serious and non-serious AEs were reported for all allocated participants who received ≥1 dose of study treatment. Per protocol, serious adverse events and all-cause mortality were collected up to 326 weeks, and non-serious adverse event data were collected up to 134 weeks.
Groups:
- Immediate Switch to MK-1439A (Day 1 to Week 24): Participants on a baseline regimen of ATRIPLA™ for at least 12 weeks prior to screening switched to blinded doravirine, tenofovir, lamivudine orally, once daily for 12 weeks, followed by open-label doravirine, tenofovir, lamivudine orally, once daily for an additional 12 weeks
- Deferred Switch to MK-1439A (Day 1 to Week 12): Participants continued their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks.
- Deferred Switch to MK-1439A (Week 12-36): Participants who continued their ongoing ATRIPLA™ regimen orally, once daily for 12 weeks switched to open-label doravirine, tenofovir, lamivudine orally, once daily for a total of 24 weeks (Week 12 - Week 36).
- Immediate Switch to MK-1439A EXT 1 (Week 24-120): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 24 - Week 120)
- Deferred Switch to MK-1439A EXT 1 (Week 36-132): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 36 - Week 132)
- Immediate Switch to MK-1439A EXT 2 (Week 120-216): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 120 - Week 216)
- Deferred Switch to MK-1439A EXT 2 (Week 132-228): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 132 - Week 228)
- Immediate Switch to MK-1439A EXT 3 (Week 216-312): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 216 - Week 312)
- Deferred Switch to MK-1439A EXT 3 (Week 228-324): One doravirine, tenofovir, lamivudine taken q.d. by mouth for an additional 96 weeks (Week 228 - Week 324)
Arm/Group | Immediate Switch to MK-1439A (Day 1 to Week 24) | Deferred Switch to MK-1439A (Day 1 to Week 12) | Deferred Switch to MK-1439A (Week 12-36) | Immediate Switch to MK-1439A EXT 1 (Week 24-120) | Deferred Switch to MK-1439A EXT 1 (Week 36-132) | Immediate Switch to MK-1439A EXT 2 (Week 120-216) | Deferred Switch to MK-1439A EXT 2 (Week 132-228) | Immediate Switch to MK-1439A EXT 3 (Week 216-312) | Deferred Switch to MK-1439A EXT 3 (Week 228-324)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/42 | 0/43 | 0/41 | 0/39 | 0/33 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 1/42 | 6/43 | 2/41 | 3/39 | 1/33 | 2/17 | 0/19
Other Adverse Events (participants affected / at risk) | 29/43 | 25/43 | 26/42 | 31/43 | 33/41 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Switch to MK-1439A (Day 1 to Week 24) (N=43) | Deferred Switch to MK-1439A (Day 1 to Week 12) (N=43) | Deferred Switch to MK-1439A (Week 12-36) (N=42) | Immediate Switch to MK-1439A EXT 1 (Week 24-120) (N=43) | Deferred Switch to MK-1439A EXT 1 (Week 36-132) (N=41) | Immediate Switch to MK-1439A EXT 2 (Week 120-216) (N=39) | Deferred Switch to MK-1439A EXT 2 (Week 132-228) (N=33) | Immediate Switch to MK-1439A EXT 3 (Week 216-312) (N=17) | Deferred Switch to MK-1439A EXT 3 (Week 228-324) (N=19)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Switch to MK-1439A (Day 1 to Week 24) (N=43) | Deferred Switch to MK-1439A (Day 1 to Week 12) (N=43) | Deferred Switch to MK-1439A (Week 12-36) (N=42) | Immediate Switch to MK-1439A EXT 1 (Week 24-120) (N=43) | Deferred Switch to MK-1439A EXT 1 (Week 36-132) (N=41) | Immediate Switch to MK-1439A EXT 2 (Week 120-216) (N=0) | Deferred Switch to MK-1439A EXT 2 (Week 132-228) (N=0) | Immediate Switch to MK-1439A EXT 3 (Week 216-312) (N=0) | Deferred Switch to MK-1439A EXT 3 (Week 228-324) (N=0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 4 (5) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 6 (6) | 2 (2) | 4 (5) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 3 (4) | 4 (4) | 4 (4) | 4 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 5 (5) | 5 (5) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (13) | 7 (9) | 3 (3) | 8 (8) | 14 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 6 (8) | 3 (3) | 5 (5) | 9 (9) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 5 (5) | 3 (3) | 3 (3) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 3 (4) | 2 (2) | 2 (2) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (2) | 7 (7) | 7 (7) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 6 (6) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 4 (4) | 5 (7) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (9) | 7 (10) | 6 (6) | 5 (5) | 10 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT02652260/Prot_SAP_001.pdf